CLINICAL TRIAL: NCT05782387
Title: A New Retrospective Natural History Study of Mucolipidosis Type IV
Brief Title: Mucolipidosis Type IV Natural History Study
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Patricia Musolino, MD PhD, Dr. Patricia Musolino, MD PhD, Massachusetts General Hospital
Other Study IDs: 2021P003131
Record Dates: First submitted 2023-02-08; First posted 2023-03-23 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Mucolipidosis Type IV
MeSH Terms: conditions — Mucolipidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The primary objectives of the study are: to describe the characteristics of the current international MLIV population; to define the median age at which patients with MLIV achieve or lose developmental milestones; to define the natural history of MLIV for the Gross Motor Function Classification System (GMFCS) (Morris and Bartlett, 2004) and the MLIV specific scale and test the validity of retrospectively applying these scales to medical record data; to define the rate of visual decline in patients with MLIV.

DETAILED DESCRIPTION:
This study is a retrospective natural history study of MLIV. It involves the collection of all participants medical records prior to the date of consent.

First, the study will provide an approximate description of the international MLIV population, which could inform the feasibility and design of interventional trials. Second, the results will be used to create an MLIV specific developmental timeline (akin to the Denver Developmental Screen (Frankenburg and Dodds, 1967)) against which a patient's developmental trajectory pre- and post-treatment can be compared. Third, the study will assess the reliability and validity of the GMFCS and our MLIV specific scales when applied retrospectively. These scales could provide longitudinal, quantitative historical data on the level of function and disability in MLIV patients. The scales could be used as endpoints in future trials or provide historical context for interpretation of treatment effects. Fourth, the study will define the rate of visual decline in patients, which could be halted by gene therapy targeted to the retina. Fifth, the study will analyze the natural history of MLIV associated EEG and brain MRI abnormalities, aiming to establish biomarkers of disease progression. And finally, the study will provide baseline data on clinical measures used to monitor for gene therapy treatment side effects (inflammatory markers, liver enzyme levels, etc.) across the life span of patient with MLIV.

ELIGIBILITY:
Inclusion Criteria:

* Patient of any age or gender with a diagnosis of MLIV confirmed through 1) genetic testing and identification of homozygous MCOLN1 allele variants known to be pathogenic, or 2) clinical characteristics consistent with MLIV and one of the following: a) electron microscopy of fibroblasts or other patient cells demonstrating abnormal lysosomal accumulations consistent with MLIV, or b) elevated gastrin levels (pathognomonic for MLIV in the setting of a neurodevelopmental disorder). Potential participants or guardians must be able to provide informed consent (patient assent is not applicable to the MLIV population).

Exclusion Criteria:

* Patients will be excluded from data collection if they do not meet any of the diagnostic criteria outlined above or they and their guardians are unable to provide informed consent. It may be possible that an initial review of collected medical records by MGH research staff after consent and enrollment suggests a misdiagnosis of MLIV. In this case the subject will be excluded from the study. Research staff will contact the patient/guardians by email and schedule a telephone or teleconference meeting to discuss the decision. All medical records will be immediately destroyed upon exclusion of a participant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We expect to enroll 50 MLIV patients who are currently in communication with the ML4 Foundation. This population is comprised of male and female patients, ages 2-45. Many patients are of Ashkenazi Jewish background. These participant candidates are located nationally and internationally.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
ML4 Characteristics | Three years
  Describe the characteristics of the current international MLIV population.
Developmental Milestones | Three years
  Define the age (median and range) at which patients with MLIV achieve or lose developmental milestones.
Gross Motor Function | Three years
  Define the natural history of MLIV for the Gross Motor Function Classification System (GMFCS) (Morris and Bartlett, 2004) and our MLIV specific scale and test the validity of retrospectively applying these scales to medical record data.
Visual Decline | Three years
  Define the rate of visual decline in patients with MLIV.

SECONDARY OUTCOMES:
Iron Deficiency and Achlorhydria | Three years
  Define the natural history of iron deficiency anemia and achlorhydria in MLIV.
Brain Imaging | Three years
  Delineate the natural history of brain imaging, including MRI, and electrophysiological features in MLIV.
Clinical Labs | Three years
  Define baseline values for clinical studies or labs that may be used to monitor gene therapy side effects in future clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Musolino, MD, PHD, Principal Investigator — Neurologist
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No